CLINICAL TRIAL: NCT03956251
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of Two Different Putty Allografts
Brief Title: Ridge Preservation With Putty Allografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, Director, Graduate Periodontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19.0516
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combined Mineralized/Demineralized Putty Allograft (Experimental): Ridge preservation with a Mineralized/Demineralized Putty allograft
  Interventions: Procedure: Combined Mineralized/Demineralized Putty Allograft
- Demineralized Putty Allograft (Active Comparator): Ridge preservation with Demineralized Putty allograft
  Interventions: Procedure: Demineralized Putty Allograft

INTERVENTIONS:
Procedure: Combined Mineralized/Demineralized Putty Allograft — At time of extraction, 15 test patients will receive ridge preservation using Combined Mineralized/Demineralized Putty Allograft
  Arms: Combined Mineralized/Demineralized Putty Allograft
Procedure: Demineralized Putty Allograft — At time of extraction, 15 control patients will receive ridge preservation using Demineralized Putty Allograft
  Arms: Demineralized Putty Allograft

SUMMARY:
The study will consist of randomized controlled clinical study trial comparing the results of a demineralized putty allorgraft versus a combined mineralized/demineralized putty allograft in approximately 30 patients, 15 per group. All materials used in the study are FDA approved.

DETAILED DESCRIPTION:
Thirty patients will be treated using the principles of guided bone regeneration utilizing a full thickness flap for ridge preservation. Fifteen test patients will receive an intrasocket demineralized and mineralized combination putty allograft (MinerOss Putty, BioHorizons) covered with a regenerative tissue matrix membrane (AlloDerm GBR, BioHorizons). The positive control group of fifteen patients will receive an intrasocket demineralized putty allograft (Puros, Zimmer) covered with a regenerative tissue matrix membrane (AlloDerm GBR, BioHorizons). Approximately, four months post-surgery, a trephine core will be taken from the grafted site immediately prior to implant placement and submitted for histologic processing.

Prior to surgery, each patient will receive a diagnostic work-up including standardized radiographs (periapicals), study casts, clinical photographs, and a clinical examination to record attachment level, probing depth, recession, and mobility of teeth adjacent to the extracted sites. Customized acrylic occlusal stents will be fabricated on the study casts to serve as fixed reference guides for the measurements. Detailed oral hygiene instructions will be provided.

For histology, trephine core specimens will be evaluated to determine percent vital bone, non-vital bone, and trabecular space. Step serial sections will be taken from each longitudinally sectioned core. The sections will be stained with hematoxylin and eosin. Ten slides per patients will be prepared with at least 4 sections per slide. For each patient, 6 of 10 slides will be assessed. The mean percentage of vital and nonvital bone, and trabecular space will be determined for each patient.

Soft tissue thickness will be measured prior to the procedure. The surgical procedure will consist of a full-thickness papilla preservation flaps performed on the buccal and palatal/lingual to expose the alveolar ridge and the tooth to be extracted. Following the extraction, vertical measurements will be taken with the acrylic occlusal stent in place, and horizontal measurements with a specially designed digital caliper. Both groups will receive an intrasocket graft covered by a regenerative tissue matrix membrane. The control group will receive a demineralized putty allograft. The test group will receive a combination mineralized and demineralized putty allograft. The surgical procedures will be documented with clinical photographs of teeth and/or intraoral structures.

Post surgical management includes all patients will be seen every 2 weeks until 8 weeks post-surgery. Patients will then be seen monthly until month 4 for the final examination and trephine core collection for histological analysis and implant placement. Patients will take doxycycline 100 mg qd for two weeks, Hydrocodone/Acetaminophen 5/325mg q4-6h as needed for pain, and naproxen 375mg q12h for one week for inflammation reduction. Postoperative visits will consist of supragingival plaque removal, and oral hygiene reinforcement Any patient who develops any significant post-operative complications or adverse reaction to the materials used or shows attachment loss greater or equal to 2 mm on teeth adjacent to the experimental site will be exited from the study and will receive appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID or steroid therapy.
10. Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in horizontal width from post-extraction site to 4-month. | 0 and 16 weeks
  Horizontal post-extraction ridge measurements at the mid-defect alveolar crest and 5 mm apical taken with a caliper.

SECONDARY OUTCOMES:
Change in post extraction ridge height. | 0 and 16 weeks
  Vertical post-extraction ridge measurements from a stent.
  * Mid socket osseous crest on facial and lingual
  * Mesial and distal socket border - facial and lingual osseous crest.
Change in facial soft tissue thickness and final occlusal soft tissue thickness. | 0 and 16 weeks
  Soft tissue thickness measurements at the crest, 5mm apical, and mid-occlusal post treatment only taken with a #40 endodontic reamer.
Histologic composition. (Histologic percent vital bone, nonvital bone and trabecular space. | 16 weeks
  Obtain via trephine core

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD MSc, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics, UofL School of Dentistry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No